CLINICAL TRIAL: NCT01335360
Title: Pharmacokinetic Evaluation of Changes in Nevirapine AUC Due to Differences in Weight
Acronym: NAWS
Status: Completed | Type: Observational
Sponsor: Western University of Health Sciences (Other)
Collaborators: Jeffrey Goodman Clinic, LA Gay & Lesbian Center (Unknown)
Responsible Party: James D. Scott, PharmD, Associate Professor, Western University
Other Study IDs: WesternU
Record Dates: First submitted 2010-12-07; First posted 2011-04-14 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infection
Keywords: nevirapine; pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Levels were drawn prior to dosing, and at the following time intervals: 0.5hr, 1hr, 1.5hr, 2hr, 4hr, 6hr, 8hr, 12hr. ~10cc of blood were drawn with each sample, centrifuged, and plasma separated into 2 cryovials. Samples were then frozen at -20oC. All samples (216) weresent to Consolidated Laboratory Services for level determination by appropriate means. All samples have now been destroyed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Subjects >80kg: As above
  Interventions: Drug: Nevirapine
- Subjects <70kg: As above
  Interventions: Drug: Nevirapine
- Subjects 70-80kg: As above
  Interventions: Drug: Nevirapine

INTERVENTIONS:
Drug: Nevirapine — 200mg twice daily of nevirapine

SUMMARY:
This study would be a prospective cohort study, stratified by weight. Patients who are stable on nevirapine for at least 3 months prior to study entry, but no more than 1year will be recruited. For 1 week, subjects will take their morning dose of nevirapine in the clinic (and be observed taking it), and given their evening dose to take at home. Subjects will need to record the date and time they take their evening dose. At the end of the week, the subjects will be sequestered at the clinic for blood draws for a 12hr pharmacokinetic sampling. They will not be brought back in at 24hrs as they will need to be redosed after 12hrs. They will have Liver Function Tests (LFT's) and other labs drawn at study entry, and one month after the end of study. Pharmacokinetic levels will be analyzed using standard mathematical models, and Area Under the Curve (AUC), Maximum concentration (Cmax), and Minimum Concentration (Cmin) will be compared between groups.

DETAILED DESCRIPTION:
This will be a non-randomized, cohort study. 8 patients in each of 3 weight ranges (< 160lb, 161-200lb, > 200lb) will be recruited to participate in the study. Subjects will be HIV + patients currently on stable therapy with nevirapine (on medication for at least 3 months with minimal self-reported adherence) as part of a combination regimen for their Human Immunodeficiency Virus (HIV) infection (as prescribed by their primary care provider). Subjects are to be in good health with liver function tests will be < 2 times normal limits, measured within 1 month prior to the study period. All subjects will be male. The reasoning for this gender bias is as follows: if both genders are to be used, there should be an equal number of male and female subjects to remove any bias from the data. Since there are not enough females taking nevirapine to be able to appropriately recruit, females will be excluded.

Subjects will be asked to take their medications the night before the study period between 8:00pm and 8:30pm, and asked to abstain from alcohol for the 7 days prior to the study. On the study day, they will report to the Jeffrey Goodman Special Care Clinic at 7:30, prior to breakfast.

Subjects will randomly be divided into 4 groups during the study period. Four healthcare professionals (one physician, one family nurse practitioner, one registered nurse and one licensed vocational nurse, will be present throughout the study for catheter insertions and blood draws. IV catheters will be inserted upon arrival, with four patients (one from each group) having a time zero and receiving their study medication at each time point of 8:00, 8:05, 8:10, 8:15, 8:20, 8:25 (this is to allow for appropriate work-flow during the blood draw portion of the study. Serial blood samples will be drawn after dosing at the following times: 0.5hr, 1hr, 1.5hr, 2hr, 4hr, 6hr, 8hr, 12hr. Subjects will be allowed to eat breakfast (supplied by the study personnel) After the 1hr blood sample. Lunch and dinner will also be available for study subjects. 12hr sample, the catheters will be removed and the subjects allowed to leave (subjects will not be allowed to leave the premises with the catheter in place). Subjects will be paid $250 for their participation after the conclusion of the study.

Consolidated Laboratory Services will analyze all blood samples for nevirapine levels. AUC's and AUC comparisons will be calculated with appropriate statistical software (Systat).

Pharmacokinetic (PK) Levels:

Levels will be drawn prior to dosing, and at the following time intervals: 0.5hr, 1hr, 1.5hr, 2hr, 4hr, 6hr, 8hr, 12hr. ~10cc of blood will be drawn with each sample, centrifuged, and plasma separated into 2 cryovials. Samples will then be frozen at -20oC. All samples (216) will be sent to Consolidated Laboratory Services for level determination by appropriate means.

Safety monitoring:

A licensed physician and a licensed family nurse practitioner will be on site for the entire study. All study personnel are certified in Basic Life Support (and some in Advanced Cardiac Life Support). The clinic facilities are equipped for minor emergencies and 911 will be utilized for major emergencies.

Statistics:

AUC's will be calculated using non-linear mathematical modeling with statistical software. AUC's will be compared using appropriate statistical tests.

Evaluation of Adverse Events:

All adverse events will be recorded and treated (if necessary) on site. Adverse events not able to be treated on site will be referred to an emergency room or to their primary provider the following day (if it is not urgent).

ELIGIBILITY:
Inclusion criteria:

1. Documented HIV infection
2. 18-50yrs of age
3. Male
4. Currently on nevirapine therapy for at least 3 months
5. LFT's < 2 times normal limits within one month prior to study date
6. In good health as judged by their primary care provider or a study provider within one month of the study date
7. Willing to abstain for 1 week prior to study date
8. No active opportunistic infections within one month prior to the study date
9. Willingness to sign informed consent

Exclusion criteria:

1. Active substance abuse
2. Poor self reported adherence to nevirapine therapy
3. Chronic liver disease or active hepatitis
4. Concurrent administration of medications with a known or suspected pharmacokinetic drug interaction with nevirapine (such as …)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: HIV positive patients stable on a nevirapine containing regimen for at least 3 months
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2003-05; Primary Completion 2003-05 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Differences in AUC based on weight/BMI | 12 hours
  This study was a "snapshot" of the PK levels following ingestion, and then compared AUC to weight and BMI.

CONTACTS AND LOCATIONS:
Overall Officials: James D Scott, PharmD, Principal Investigator — Western University of Health Sciences
Locations (1):
- Jeffrey Goodman Clinic, Los Angeles, California, United States